CLINICAL TRIAL: NCT02924506
Title: Cervical Arthroplasty "Fixed Core" Versus "Movable Core": A Controlled Prospective Study, Clinical and Radiological Impact in the Medium Term
Brief Title: Cervical Arthroplasty "Fixed Core" Versus "Movable Core": Clinical and Radiological Impact in the Medium Term
Acronym: DISC-C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Moving of coordinator.
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRO-2014-04
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Neck Pain; Back Pain
Keywords: cervical arthroplasty
MeSH Terms: conditions — Neck Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Core (Other): Cervical arthroplasty with fixed core prothesis
  Interventions: Device: ProDisc-C prothesis
- Movable Core (Other): Cervical arthroplasty with movable core prothesis
  Interventions: Device: Mobi-C prothesis

INTERVENTIONS:
Device: Mobi-C prothesis — Mobi-C Prothesis, LDR Medical (company)
  Arms: Movable Core
Device: ProDisc-C prothesis — ProDisc-C prothesis, Vivo Depuy Synthes (company)
  Arms: Fixed Core

SUMMARY:
Nowadays, there is no clinical and radiological study comparing two different types of mobile implants in patients requiring surgical treatment for symptomatic cervical disc disease. Thus, the choice of the ideal implant remains uncertain.

The goal of this work is to compare the impact of two types of mobile implants in height drives, solicitation facets, positioning and collection of prostheses within the intervertebral spaces.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Symptomatic cervical disc degenerative pathologies to 1 or more contiguous or non-contiguous levels C3-4 to C6-7.
* Symptoms including: Cervicobrachial neuralgia and / or Loss of root muscle strength and / or Sensory impairment and paresthesia and / or Cervical myelopathy table
* Concordant diagnosis confirmed by CT (Computerized Tomography scanner) and MRI (Magnetic Resonance Imaging) of the cervical spine
* NPDS (Neck Pain and Disability Scale) > 30
* Failure to respond to conservative medical treatment for 6 weeks or worsening symptoms despite conservative treatment
* Physical and mental fitness to ensure compliance with the protocol
* Signed informed consent

Exclusion Criteria:

* Unstable cervical spine injuries requiring fusion C1 to C7 for whatever the etiology, proven on dynamic views of the cervical spine
* Paget's disease, osteomalacia, other metabolic bone diseases
* Chronic corticosteroid use
* Active tumor pathology
* Segmental angulation < -11 ° or > 11 ° at the respective segment or adjacent segments on static images of the cervical spine
* Known allergy to Chromium, Cobalt, Mobdylene (chemical element), Polyethylene, or Titanium
* History of surgery in the previous 30 days before inclusion
* History of mental illness or disability involving a "safeguard procedure justice of the person"
* Contraindications to non steroidal anti inflammatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Neck Pain and Disability Scale (NPDS) between the two groups | Baseline
Neck Pain and Disability Scale (NPDS) between the two groups | 3 months
Neck Pain and Disability Scale (NPDS) between the two groups | 1 year
Neck Pain and Disability Scale (NPDS) between the two groups | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DUFOUR, Ph, Principal Investigator — CHR d'Orleans
Locations (2):
- France (2):
  - CHR d'ORLEANS, Orléans
  - Hôpital Bretonneau, CHU DE TOURS, Tours

IPD SHARING:
Plan to Share IPD: No